CLINICAL TRIAL: NCT05743621
Title: A Phase I, Open-Label, Dose-Finding Study of TVB-2640 Administered in Combination With Enzalutamide (Xtandi) in Men With Metastatic Castration-Resistant Prostate Cancer (mCRPC)
Brief Title: Study of TVB-2640 in Men With Metastatic Castration-Resistant Prostate Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Sagimet Biosciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-08025117
Record Dates: First submitted 2023-01-30; First posted 2023-02-24 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Prostatic Neoplasms, Castration-Resistant
Keywords: Metastatic Castration-Resistant Prostate Cancer; FASN Inhibitor
MeSH Terms: conditions — Prostatic Neoplasms, Castration-Resistant | interventions — TVB-2640; enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TVB-2640 in combination with Enzalutamide (Experimental)
  Interventions: Drug: TVB-2640; Drug: Enzalutamide

INTERVENTIONS:
Drug: TVB-2640 — TVB- 2640 at 100 mg, 150mg, 200 mg, 250 mg, or 300mg daily, orally; dose determined by BOIN dose escalation per the protocol
Drug: Enzalutamide — 160 mg daily PO
  Other Names: Xtandi

SUMMARY:
The purpose of this study is to determine what effects (good and bad) Enzalutamide and TVB-2640 have in the treatment of prostate cancer whose prostate cancer has spread to other parts of their body and that has not gotten better with previous treatment. This study is a Phase I clinical trial. Phase I clinical trials test the side effects of an investigational drug or an investigational combination with another drug. "Investigational" means that the drug is still being studied and research doctors are trying to find out more about it. Although Enzalutamide is already being used to treat men with prostate cancer, combining Enzalutamide with TVB-2640 together in patients with prostate cancer is considered experimental. This research study is being done because additional effective treatments are needed for prostate cancer that has spread and is growing despite hormone suppression. By doing this study, the investigators hope to learn if combining Enzalutamide with TVB-2640 can be done safely. Participation in this research will last about 12 to 24 months after enrollment.

DETAILED DESCRIPTION:
This phase I, open-label, dose-escalation study is designed to evaluate the dose limiting toxicities (DLTs) and maximum-tolerated dose (MTD) of TVB-2640 plus Enzalutamide and establish the TVB-2640 dose recommended for further investigation in phase 2 (i.e., recommended phase 2 dose [RP2D]). Patients with a confirmed histological or cytological diagnosis of prostate cancer (PC), evidence of metastatic PC on imaging (bone scan and/or CT/MRI scan), serum testosterone <50 ng/dl, who had progressed on androgen-depletion therapy (ADT), with documented progressive metastatic castration-resistant prostate cancer (mCRPC) based on Prostate Cancer Working Group 3 (PCWG3) criteria and no previously treatment with cytotoxic chemotherapy are eligible. This study represents the first clinical evaluation of TVB-2640 in combination with Enzalutamide. All patients will receive Enzalutamide monotherapy at the approved dose of 160 mg once daily for 28 days to reach the steady state as determined by measuring Enzalutamide and des-methyl-Enzalutamide levels. Participants who complete the Enzalutamide run-in period will begin oral TVB-2640 at the dose of 100 mg. The dose escalation scheme will be the Bayesian optimal interval (BOIN) design with additional dose levels of 100 mg, 150mg, 200 mg, 250 mg, and 300mg daily. The maximum sample size for the phase I will be 30 patients and the target DLT rate is 25% or less and a maximum of 9 patients at any dose level.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Documented histological or cytological diagnosis of PC
* Evidence of metastatic PC on imaging (bone scan and/or CT/MRI scan)
* Diagnosis of progressive metastatic, castration resistant prostate cancer
* Potential participant must be planning to receive Enzalutamide as their first line of therapy for castration resistant prostate cancer or have previously received up to one line of Abiraterone or an androgen receptor antagonist
* Willing to undergo a tumor biopsy prior to beginning therapy, if recent tissue samples are not available
* Willing to undergo a tumor biopsy of at least one metastatic site or primary prostate after ~4-6 weeks of therapy with both agents
* Participants without prior orchiectomy must be currently taking and willing to continue luteinizing hormone-releasing hormone (LHRH) analogue (agonist or antagonist) therapy until permanent discontinuation of study treatment
* ECOG performance status of 0-1
* Recovery to baseline or ≤ Grade 1 CTCAE v5 from toxicities related to any prior treatments, unless specified below AE(s) are clinically nonsignificant and/or stable on supportive therapy
* Adequate organ and marrow function, based upon laboratory criteria within 14 days before first dose of study treatment
* Sexually active, fertile participants and their partners must agree to use medically accepted methods of contraception (e.g., barrier methods, including male condom with spermicide during the course of the study and for 4 months after the last dose of study treatment
* Capable of understanding and complying with the protocol requirements and must have signed the informed consent document

Exclusion Criteria:

* Receipt of any type of biologic, or other systemic anticancer therapy (including investigational) except agents within 4 weeks before first dose of study treatment. Anti-resorptive bone agents are also allowed.
* Radiation therapy for bone metastasis within 2 weeks, any other radiation therapy within 4 weeks before first dose of study treatment. Systemic treatment with radionuclides within 6 weeks before the first dose of study treatment. Participants with clinically relevant ongoing complications from prior radiation therapy are not eligible.
* Prior exposure to taxane chemotherapy
* History of pneumonitis
* Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery (including radiosurgery) and stable for at least 4 weeks prior to first dose of study treatment after radiotherapy or at least 4 weeks prior to first dose of study treatment after major surgery (e.g., removal or biopsy of brain metastasis). Participants must have complete wound healing from major surgery or minor surgery before first dose of study treatment. Eligible participants must be neurologically asymptomatic and without corticosteroid treatment for neurological indications at the time of first dose of study treatment.
* Participants with clinically significant dry eye or corneal abnormalities
* Currently taking certain anticoagulation medications, such as coumarin agents (e.g., warfarin), direct thrombin inhibitors (e.g., dabigatran), direct factor Xa inhibitor betrixaban, or platelet inhibitors (e.g., clopidogrel)
* Participant has prothrombin time (PT)/INR or partial thromboplastin time (PTT) test ≥ 1.3 X the laboratory ULN within 30 days before the first dose of study treatment.
* Participants should not receive strong CYP2C8 or strong P-gp inhibitors; strong CYP3A4 or CYP2C8 inducers; and strong CYP3A4, CYP2C9 and CYP2C19 substrates while participating in the trial, unless utilized with caution to treat a drug-related AE when no alternative is available and discussed with the Medical Monitor.
* Participant has uncontrolled, significant intercurrent or recent Cardiovascular disorders including, but not limited to, the following conditions:

  i. Congestive heart failure New York Heart Association Class 3 or 4, unstable angina pectoris, serious cardiac arrhythmias.

ii. Uncontrolled hypertension defined as sustained blood pressure (BP) >140 mm Hg systolic or >90 mm Hg diastolic despite optimal antihypertensive treatment.

iii. Stroke (including transient ischemic attack [TIA]), myocardial infarction (MI), or other ischemic event, or thromboembolic event (e.g. deep venous thrombosis, pulmonary embolism) within 6 months before first dose.

* Corrected QT interval calculated by the Fridericia formula (QTcF) > 470 ms per electrocardiogram (ECG) within 28 days before first dose of study treatment.
* Inability to swallow tablets.
* Use of herbal products that may decrease PSA levels within 4 weeks prior to enrollment
* Previously identified allergy or hypersensitivity to components of the study treatment formulations.
* Diagnosis of another type of cancer within 2 years before first dose of study treatment, except for superficial skin cancers, or localized, low-grade tumors deemed cured and not treated with systemic therapy.
* Any serious and/or unstable pre-existing medical, psychiatric disorder or other conditions that could interfere with participant's safety, obtaining informed consent or compliance to the study procedures.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-11-20 (Actual); Primary Completion 2027-01-25 (Estimated); Study Completion 2029-01-25 (Estimated)

PRIMARY OUTCOMES:
Optimal dose of TVB-2640 in combination with Enzalutamide, as determined by the maximum tolerated dose (MTD) | Day 28
  The maximum tolerated dose (MTD) is defined as the highest dose level at which ≤1 patient experiences a dose-limiting toxicity, as defined in the protocol (DLT). Once all the patients are accrued, the MTD will be determined by performing isotonic regression on the pooled data.

SECONDARY OUTCOMES:
Number of adverse events (evaluated using the NCI CTCAE v5.0) of different doses of TVB-2640 in combination with Enzalutamide | 12 months
  All observed AEs will be tabulated and reported as relative frequencies (i.e., fraction of patients with that AE). This will be done by AE and maximum grade experienced within a patient. The fraction of patients with each AE by grade will be estimated with a binomial point estimate and corresponding 95% binomial confidence interval (CI). AEs will be collected until 30 days following the last dose of study drug. AEs will be reported for each different dose of TVB-2640 given.
Mean TVB-2640 total exposure (as measured by the area under the drug serum concentration vs. the time from administration curve [AUC]) | Day 28; Days 36-37; Days 43-44; Days 50-51
  Peripheral blood will be drawn at:
  Day 28:
  * Pre- enza dose
  * Post-dose
  * 1 hours (±5 min)
  * 2 hours (±5 min)
  * 4 hours (±30 min)
  Days 36-37:
  * Pre-TVB-2640 dose
  * Post-dose
  * 2 hours (±5 min)
  * 4 hours (±30 min)
  * 6 hours (±30 min)
  * 8 hours (±30 min)
  * 24-hours (±1 hour)
  Days 43-44:
  * Pre-TVB-2640 dose
  * Post-dose
  * 30 minutes (±5 min)
  * 1 hour (±5 min)
  * 2 hours (±5 min)
  * 4 hours (±30 min)
  * 6 hours (±30 min)
  * 8 hours (±30 min)
  * 24-hours (±1 hour)
  Days 50-51:
  * Pre-TVB-2640 dose
  * Post-dose
  * 30 minutes (±5 min)
  * 1 hour (±5 min)
  * 2 hours (±5 min)
  * 4 hours (±30 min)
  * 6 hours (±30 min)
  * 8 hours (±30 min)
  * 24-hours (±1 hour)
Mean Enzalutamide total exposure (as measured by the area under the drug serum concentration vs. the time from administration curve [AUC]) | Day 28; Days 36-37; Days 43-44; Days 50-51
  Peripheral blood will be drawn at:
  Day 28:
  * Pre- enza dose
  * Post-dose
  * 1 hours (±5 min)
  * 2 hours (±5 min)
  * 4 hours (±30 min)
  Days 36-37:
  * Pre-TVB-2640 dose
  * Post-dose
  * 2 hours (±5 min)
  * 4 hours (±30 min)
  * 6 hours (±30 min)
  * 8 hours (±30 min)
  * 24-hours (±1 hour)
  Days 43-44:
  * Pre-TVB-2640 dose
  * Post-dose
  * 30 minutes (±5 min)
  * 1 hour (±5 min)
  * 2 hours (±5 min)
  * 4 hours (±30 min)
  * 6 hours (±30 min)
  * 8 hours (±30 min)
  * 24-hours (±1 hour)
  Days 50-51:
  * Pre-TVB-2640 dose
  * Post-dose
  * 30 minutes (±5 min)
  * 1 hour (±5 min)
  * 2 hours (±5 min)
  * 4 hours (±30 min)
  * 6 hours (±30 min)
  * 8 hours (±30 min)
  * 24-hours (±1 hour)
Mean maximum serum concentration (Cmax) of TVB-2640 | Day 28; Days 36-37; Days 43-44; Days 50-51
  Peripheral blood will be drawn at the following times:
  Day 28:
  * Pre- enza dose
  * 1 hours (±5 min) post-dose
  * 2 hours (±5 min) post-dose
  * 4 hours (±30 min) post-dose
  Days 36-37:
  * Before TVB-2640 administration
  * 2 hours (±5 min) post-dose
  * 4 hours (±30 min) post-dose
  * 6 hours (±30 min) post-dose
  * 8 hours (±30 min) post-dose
  * 24-hours (±1 hour) post-dose
  Days 43-44:
  * Before TVB-2640 administration
  * 30 minutes (±5 min) post-dose
  * 1 hour (±5 min) post-dose
  * 2 hours (±5 min) post-dose
  * 4 hours (±30 min) post-dose
  * 6 hours (±30 min) post-dose
  * 8 hours (±30 min) post-dose
  * 24-hours (±1 hour) post-dose
  Days 50-51:
  * Before TVB-2640 administration
  * 30 minutes (±5 min) post-dose
  * 1 hour (±5 min) post-dose
  * 2 hours (±5 min) post-dose
  * 4 hours (±30 min) post-dose
  * 6 hours (±30 min) post-dose
  * 8 hours (±30 min) post-dose
  * 24-hours (±1 hour) post-dose
Mean maximum serum concentration (Cmax) of Enzalutamide | Day 28; Days 36-37; Days 43-44; Days 50-51
  Peripheral blood will be drawn at the following times:
  Day 28:
  * Pre- enza dose
  * 1 hours (±5 min) post-dose
  * 2 hours (±5 min) post-dose
  * 4 hours (±30 min) post-dose
  Days 36-37:
  * Before TVB-2640 administration
  * 2 hours (±5 min) post-dose
  * 4 hours (±30 min) post-dose
  * 6 hours (±30 min) post-dose
  * 8 hours (±30 min) post-dose
  * 24-hours (±1 hour) post-dose
  Days 43-44:
  * Before TVB-2640 administration
  * 30 minutes (±5 min) post-dose
  * 1 hour (±5 min) post-dose
  * 2 hours (±5 min) post-dose
  * 4 hours (±30 min) post-dose
  * 6 hours (±30 min) post-dose
  * 8 hours (±30 min) post-dose
  * 24-hours (±1 hour) post-dose
  Days 50-51:
  * Before TVB-2640 administration
  * 30 minutes (±5 min) post-dose
  * 1 hour (±5 min) post-dose
  * 2 hours (±5 min) post-dose
  * 4 hours (±30 min) post-dose
  * 6 hours (±30 min) post-dose
  * 8 hours (±30 min) post-dose
  * 24-hours (±1 hour) post-dose
Mean minimum serum concentration (Cmin) of TVB-2640 | Day 28; Days 36-37; Days 43-44; Days 50-51
  Peripheral blood will be drawn at the following times:
  Day 28:
  * Pre- enza dose
  * 1 hours (±5 min) post-dose
  * 2 hours (±5 min) post-dose
  * 4 hours (±30 min) post-dose
  Days 36-37:
  * Before TVB-2640 administration
  * 2 hours (±5 min) post-dose
  * 4 hours (±30 min) post-dose
  * 6 hours (±30 min) post-dose
  * 8 hours (±30 min) post-dose
  * 24-hours (±1 hour) post-dose
  Days 43-44:
  * Before TVB-2640 administration
  * 30 minutes (±5 min) post-dose
  * 1 hour (±5 min) post-dose
  * 2 hours (±5 min) post-dose
  * 4 hours (±30 min) post-dose
  * 6 hours (±30 min) post-dose
  * 8 hours (±30 min) post-dose
  * 24-hours (±1 hour) post-dose
  Days 50-51:
  * Before TVB-2640 administration
  * 30 minutes (±5 min) post-dose
  * 1 hour (±5 min) post-dose
  * 2 hours (±5 min) post-dose
  * 4 hours (±30 min) post-dose
  * 6 hours (±30 min) post-dose
  * 8 hours (±30 min) post-dose
  * 24-hours (±1 hour) post-dose
Mean minimum serum concentration (Cmin) of Enzalutamide | Day 28; Days 36-37; Days 43-44; Days 50-51
  Peripheral blood will be drawn at the following times:
  Day 28:
  * Pre- enza dose
  * 1 hours (±5 min) post-dose
  * 2 hours (±5 min) post-dose
  * 4 hours (±30 min) post-dose
  Days 36-37:
  * Before TVB-2640 administration
  * 2 hours (±5 min) post-dose
  * 4 hours (±30 min) post-dose
  * 6 hours (±30 min) post-dose
  * 8 hours (±30 min) post-dose
  * 24-hours (±1 hour) post-dose
  Days 43-44:
  * Before TVB-2640 administration
  * 30 minutes (±5 min) post-dose
  * 1 hour (±5 min) post-dose
  * 2 hours (±5 min) post-dose
  * 4 hours (±30 min) post-dose
  * 6 hours (±30 min) post-dose
  * 8 hours (±30 min) post-dose
  * 24-hours (±1 hour) post-dose
  Days 50-51:
  * Before TVB-2640 administration
  * 30 minutes (±5 min) post-dose
  * 1 hour (±5 min) post-dose
  * 2 hours (±5 min) post-dose
  * 4 hours (±30 min) post-dose
  * 6 hours (±30 min) post-dose
  * 8 hours (±30 min) post-dose
  * 24-hours (±1 hour) post-dose
Mean TVB-2640 volume of distribution at steady state | Day 28; Days 36-37; Days 43-44; Days 50-51
  Peripheral blood will be drawn at the following times:
  Day 28:
  * Pre- enza dose
  * 1 hours (±5 min) post-dose
  * 2 hours (±5 min) post-dose
  * 4 hours (±30 min) post-dose
  Days 36-37:
  * Before TVB-2640 administration
  * 2 hours (±5 min) post-dose
  * 4 hours (±30 min) post-dose
  * 6 hours (±30 min) post-dose
  * 8 hours (±30 min) post-dose
  * 24-hours (±1 hour) post-dose
  Days 43-44:
  * Before TVB-2640 administration
  * 30 minutes (±5 min) post-dose
  * 1 hour (±5 min) post-dose
  * 2 hours (±5 min) post-dose
  * 4 hours (±30 min) post-dose
  * 6 hours (±30 min) post-dose
  * 8 hours (±30 min) post-dose
  * 24-hours (±1 hour) post-dose
  Days 50-51:
  * Before TVB-2640 administration
  * 30 minutes (±5 min) post-dose
  * 1 hour (±5 min) post-dose
  * 2 hours (±5 min) post-dose
  * 4 hours (±30 min) post-dose
  * 6 hours (±30 min) post-dose
  * 8 hours (±30 min) post-dose
  * 24-hours (±1 hour) post-dose
Mean Enzalutamide volume of distribution at steady state | Day 28; Days 36-37; Days 43-44; Days 50-51
  Peripheral blood will be drawn at the following times:
  Day 28:
  * Pre- enza dose
  * 1 hours (±5 min) post-dose
  * 2 hours (±5 min) post-dose
  * 4 hours (±30 min) post-dose
  Days 36-37:
  * Before TVB-2640 administration
  * 2 hours (±5 min) post-dose
  * 4 hours (±30 min) post-dose
  * 6 hours (±30 min) post-dose
  * 8 hours (±30 min) post-dose
  * 24-hours (±1 hour) post-dose
  Days 43-44:
  * Before TVB-2640 administration
  * 30 minutes (±5 min) post-dose
  * 1 hour (±5 min) post-dose
  * 2 hours (±5 min) post-dose
  * 4 hours (±30 min) post-dose
  * 6 hours (±30 min) post-dose
  * 8 hours (±30 min) post-dose
  * 24-hours (±1 hour) post-dose
  Days 50-51:
  * Before TVB-2640 administration
  * 30 minutes (±5 min) post-dose
  * 1 hour (±5 min) post-dose
  * 2 hours (±5 min) post-dose
  * 4 hours (±30 min) post-dose
  * 6 hours (±30 min) post-dose
  * 8 hours (±30 min) post-dose
  * 24-hours (±1 hour) post-dose
Mean time to maximum TVB-2640 serum concentration (Tmax) after administration | Day 28; Days 36-37; Days 43-44; Days 50-51
  Peripheral blood will be drawn at the following times:
  Day 28:
  * Pre- enza dose
  * 1 hours (±5 min) post-dose
  * 2 hours (±5 min) post-dose
  * 4 hours (±30 min) post-dose
  Days 36-37:
  * Before TVB-2640 administration
  * 2 hours (±5 min) post-dose
  * 4 hours (±30 min) post-dose
  * 6 hours (±30 min) post-dose
  * 8 hours (±30 min) post-dose
  * 24-hours (±1 hour) post-dose
  Days 43-44:
  * Before TVB-2640 administration
  * 30 minutes (±5 min) post-dose
  * 1 hour (±5 min) post-dose
  * 2 hours (±5 min) post-dose
  * 4 hours (±30 min) post-dose
  * 6 hours (±30 min) post-dose
  * 8 hours (±30 min) post-dose
  * 24-hours (±1 hour) post-dose
  Days 50-51:
  * Before TVB-2640 administration
  * 30 minutes (±5 min) post-dose
  * 1 hour (±5 min) post-dose
  * 2 hours (±5 min) post-dose
  * 4 hours (±30 min) post-dose
  * 6 hours (±30 min) post-dose
  * 8 hours (±30 min) post-dose
  * 24-hours (±1 hour) post-dose
Mean time to maximum Enzalutamide serum concentration (Tmax) after administration | Day 28; Days 36-37; Days 43-44; Days 50-51
  Peripheral blood will be drawn at the following times:
  Day 28:
  * Pre- enza dose
  * 1 hours (±5 min) post-dose
  * 2 hours (±5 min) post-dose
  * 4 hours (±30 min) post-dose
  Days 36-37:
  * Before TVB-2640 administration
  * 2 hours (±5 min) post-dose
  * 4 hours (±30 min) post-dose
  * 6 hours (±30 min) post-dose
  * 8 hours (±30 min) post-dose
  * 24-hours (±1 hour) post-dose
  Days 43-44:
  * Before TVB-2640 administration
  * 30 minutes (±5 min) post-dose
  * 1 hour (±5 min) post-dose
  * 2 hours (±5 min) post-dose
  * 4 hours (±30 min) post-dose
  * 6 hours (±30 min) post-dose
  * 8 hours (±30 min) post-dose
  * 24-hours (±1 hour) post-dose
  Days 50-51:
  * Before TVB-2640 administration
  * 30 minutes (±5 min) post-dose
  * 1 hour (±5 min) post-dose
  * 2 hours (±5 min) post-dose
  * 4 hours (±30 min) post-dose
  * 6 hours (±30 min) post-dose
  * 8 hours (±30 min) post-dose
  * 24-hours (±1 hour) post-dose
Mean Serum half-life (T1/2) of TVB-2640 | Day 28; Days 36-37; Days 43-44; Days 50-51
  Peripheral blood will be drawn at the following times:
  Day 28:
  * Pre- enza dose
  * 1 hours (±5 min) post-dose
  * 2 hours (±5 min) post-dose
  * 4 hours (±30 min) post-dose
  Days 36-37:
  * Before TVB-2640 administration
  * 2 hours (±5 min) post-dose
  * 4 hours (±30 min) post-dose
  * 6 hours (±30 min) post-dose
  * 8 hours (±30 min) post-dose
  * 24-hours (±1 hour) post-dose
  Days 43-44:
  * Before TVB-2640 administration
  * 30 minutes (±5 min) post-dose
  * 1 hour (±5 min) post-dose
  * 2 hours (±5 min) post-dose
  * 4 hours (±30 min) post-dose
  * 6 hours (±30 min) post-dose
  * 8 hours (±30 min) post-dose
  * 24-hours (±1 hour) post-dose
  Days 50-51:
  * Before TVB-2640 administration
  * 30 minutes (±5 min) post-dose
  * 1 hour (±5 min) post-dose
  * 2 hours (±5 min) post-dose
  * 4 hours (±30 min) post-dose
  * 6 hours (±30 min) post-dose
  * 8 hours (±30 min) post-dose
  * 24-hours (±1 hour) post-dose
Mean Serum half-life (T1/2) of Enzalutamide | Day 28; Days 36-37; Days 43-44; Days 50-51
  Peripheral blood will be drawn at the following times:
  Day 28:
  * Pre- enza dose
  * 1 hours (±5 min) post-dose
  * 2 hours (±5 min) post-dose
  * 4 hours (±30 min) post-dose
  Days 36-37:
  * Before TVB-2640 administration
  * 2 hours (±5 min) post-dose
  * 4 hours (±30 min) post-dose
  * 6 hours (±30 min) post-dose
  * 8 hours (±30 min) post-dose
  * 24-hours (±1 hour) post-dose
  Days 43-44:
  * Before TVB-2640 administration
  * 30 minutes (±5 min) post-dose
  * 1 hour (±5 min) post-dose
  * 2 hours (±5 min) post-dose
  * 4 hours (±30 min) post-dose
  * 6 hours (±30 min) post-dose
  * 8 hours (±30 min) post-dose
  * 24-hours (±1 hour) post-dose
  Days 50-51:
  * Before TVB-2640 administration
  * 30 minutes (±5 min) post-dose
  * 1 hour (±5 min) post-dose
  * 2 hours (±5 min) post-dose
  * 4 hours (±30 min) post-dose
  * 6 hours (±30 min) post-dose
  * 8 hours (±30 min) post-dose
  * 24-hours (±1 hour) post-dose
Mean TVB-2640 clearance | Day 28; Days 36-37; Days 43-44; Days 50-51
  Peripheral blood will be drawn at the following times:
  Day 28:
  * Pre- enza dose
  * 1 hours (±5 min) post-dose
  * 2 hours (±5 min) post-dose
  * 4 hours (±30 min) post-dose
  Days 36-37:
  * Before TVB-2640 administration
  * 2 hours (±5 min) post-dose
  * 4 hours (±30 min) post-dose
  * 6 hours (±30 min) post-dose
  * 8 hours (±30 min) post-dose
  * 24-hours (±1 hour) post-dose
  Days 43-44:
  * Before TVB-2640 administration
  * 30 minutes (±5 min) post-dose
  * 1 hour (±5 min) post-dose
  * 2 hours (±5 min) post-dose
  * 4 hours (±30 min) post-dose
  * 6 hours (±30 min) post-dose
  * 8 hours (±30 min) post-dose
  * 24-hours (±1 hour) post-dose
  Days 50-51:
  * Before TVB-2640 administration
  * 30 minutes (±5 min) post-dose
  * 1 hour (±5 min) post-dose
  * 2 hours (±5 min) post-dose
  * 4 hours (±30 min) post-dose
  * 6 hours (±30 min) post-dose
  * 8 hours (±30 min) post-dose
  * 24-hours (±1 hour) post-dose
Mean Enzalutamide clearance | Day 28; Days 36-37; Days 43-44; Days 50-51
  Peripheral blood will be drawn at the following times:
  Day 28:
  * Pre- enza dose
  * 1 hours (±5 min) post-dose
  * 2 hours (±5 min) post-dose
  * 4 hours (±30 min) post-dose
  Days 36-37:
  * Before TVB-2640 administration
  * 2 hours (±5 min) post-dose
  * 4 hours (±30 min) post-dose
  * 6 hours (±30 min) post-dose
  * 8 hours (±30 min) post-dose
  * 24-hours (±1 hour) post-dose
  Days 43-44:
  * Before TVB-2640 administration
  * 30 minutes (±5 min) post-dose
  * 1 hour (±5 min) post-dose
  * 2 hours (±5 min) post-dose
  * 4 hours (±30 min) post-dose
  * 6 hours (±30 min) post-dose
  * 8 hours (±30 min) post-dose
  * 24-hours (±1 hour) post-dose
  Days 50-51:
  * Before TVB-2640 administration
  * 30 minutes (±5 min) post-dose
  * 1 hour (±5 min) post-dose
  * 2 hours (±5 min) post-dose
  * 4 hours (±30 min) post-dose
  * 6 hours (±30 min) post-dose
  * 8 hours (±30 min) post-dose
  * 24-hours (±1 hour) post-dose
Prostate-Specific Antigen (PSA) Response Rate | Baseline; 12 weeks
  The PSA response rate will be evaluated using PCWG3 criteria and defined as the proportion of patients with a PSA decline of at least 50%. Any change from baseline is confirmed by a second measurement at least 3 weeks later. PSA Response Rate will be evaluated using PCWG3 criteria and defined as following: Percentage change from baseline in PSA to 12 weeks post Enzalutamide plus TVB-2640. Only evaluate for patients with at least 12 weeks of treatment, the PSA assessment at 12 weeks (84 days +/-3 days) will be used; Maximum percent decrease in PSA from baseline that occurs at any point after treatment.
Overall radiographic response rate | From baseline until disease progression for a maximum of 2 years from enrollment
  Tumor response will be evaluated using the PCWG3 criteria. Patients with measurable disease will be evaluated for clinical benefit as determined by tumor response using RECIST v1.1. Patients with non-measurable bone disease will be evaluated for progression based on the presence of any new lesions by bone scans. Radiographic tumor evaluation will be performed at screening and every 3 cycles or more frequently as determined by the investigator. Using the tumor response that is determined by the investigator, best overall response will be determined using RECIST v1.1. Best overall response is defined as the best response recorded from the start of treatment until disease progression or study exit. The overall response rate will be determined as the number of patients with a confirmed PR or CR divided by the total number of patients evaluable for overall response.
Overall median progression free survival (PFS) | From baseline until disease progression or death from any cause for a maximum of 2 years from enrollment
  Overall progression free survival (PFS) is determined using the PCWG3 criteria. Overall PFS is measured from screening until the time that disease progression (radiographic progressive disease or clinical deterioration) or death is documented, whichever occurs first.
Median radiographic progression free survival (PFS) as assessed by PCWG3 | From baseline until disease progression for a maximum of 2 years from enrollment
  Radiographic progression-free survival (rPFS) is determined using the PCWG3 criteria to assess both soft-tissue and bone assessments. The rPFS is measured from screening until the time the first radiographic scan shows disease progression, or until the time of death, whichever occurs first. Patients who do not progress radiographically or did not die prior to study exit are censored on the date of their last dose of Enzalutamide plus TVB-2640. PFS will be summarized with a Kaplan-Meier curve. The Kaplan-Meier estimator will be used to determine the 6-month and 12-month PFS rates. Each estimate will have a corresponding 95% confidence interval. The median PFS will also be estimated with a corresponding 95% confidence interval

CONTACTS AND LOCATIONS:
Overall Officials: David Nanus, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine/NewYork-Presbyterian Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No